CLINICAL TRIAL: NCT06067646
Title: From Guidelines to Clinical Care: What is Needed for Optimizing Counceling on Feeding Options of Babies From Mothers Living With HIV?
Brief Title: Optimizing Counceling on Feeding Options of Babies From Mothers Living With HIV
Acronym: ROMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-16739
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health care providers involved in care for people living with hiv (Other): Semi-structured interviews with health care providers
  Interventions: Behavioral: Semistructured interview
- People living with HIV with prior pregnancy or desire to have children (Other): Semi-structured interviews with people living with HIV with prior pregnancy or desire to have children
  Interventions: Behavioral: Semistructured interview

INTERVENTIONS:
Behavioral: Semistructured interview — Semistructured interview and validated quality of life assesment using EQ5-DL

SUMMARY:
Semi structured interviews will be performed to determine attitudes and experiences of people living with HIV and health care providers on counseling on feeding options of babies from mothers living with HIV in order to optimize counseling in the future

ELIGIBILITY:
Inclusion Criteria:

* Health care provider involved in care for people living with HIV in Duth HIV treatment facility or
* Person living with HIV + age 18-45 + prior pregnancy/desire to have children

Exclusion Criteria:

* Insufficient command of Dutch or English language (oral)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Experiences and attitudes on subject | Explore during semistructured interview during 1 to 2 hours
  Experiences and attitudes on subject

CONTACTS AND LOCATIONS:
Overall Officials: Angela Colbers, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No